CLINICAL TRIAL: NCT06703138
Title: Role of MRI Diffusion in Differentiation Between Various Vertebral Bone Marrow Pathological Lesions. .
Brief Title: Role of Diffusion MRI in Differentiation of Various Bone Marrow Lesions
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zainab Hassan Mahmoud Nafadi, Principal Investigator, Assiut University
Other Study IDs: MRI in bone marrow lesions
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Diffusion MRI; Bone Marrow Disease
Keywords: MRI; Bone marrow pathologies
MeSH Terms: conditions — Bone Marrow Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bone marrow lesions are common, and imaging findings are associated with various aetiologies, as compared to conventional radiography and computed tomography (CT), MRI is a better non-invasive imaging modality to evaluate vertebral bone marrow, due to better soft-tissue contrast, so the aim of our study is the use of MRI diffusion in differentiating various vertebral bone marrow pathological lesions.

DETAILED DESCRIPTION:
Bone marrow lesions are common, and imaging findings are associated with various aetiologies, such as degenerative, infectious, traumatic, malignant, metabolic, and haematopoietic .

As compared to conventional radiography and computed tomography (CT), MRI is a better non-invasive imaging modality to evaluate vertebral bone marrow, due to better soft-tissue contrast as well as being non-ionising in nature .

Although conventional MRI is essential for anatomical visualization and lesion detection in bone marrow pathologies ,but it often insufficient in distinguishing different vertebral bone marrow lesions, due to overlapping imaging features and often due to coexistence of bone marrow oedema that can be caused by fractures, infection, and bone marrow hyperplasia, thus reducing the specificity of conventional sequences .

MRI diffusion provides complementary information about tissue microstructure and cellular .it exploits the translational mobility of water molecules to obtain information on the microscopic behaviour of the tissues.

On the other hand, apparent diffusion coefficient (ADC) values provide quantitative measure of Brownian movement with low ADC values implying restricted diffusion and high values being a measure of free diffusion.

Therefore, DWI provides both qualitative and quantitative functional information concerning the microscopic movements of water at the cellular level. The benefits of DWI comprise a small scanning period that allows it to be easily included in the routine imaging protocols .

For example, In healthy bone marrow, water diffusion is relatively unrestricted due to its cellularity and vascularity, while pathologies such as metastatic disease or myelofibrosis typically exhibit restricted diffusion.

Diffusion MRI can also distinguish bone marrow edema like acute injury or inflammation, from infiltrative diseases such as multiple myeloma. Edema typically shows higher ADC values due to the increased water content, whereas infiltrative diseases reduce diffusion, resulting in lower ADC values.

These examples illustrate how MRI diffusion can differentiate various vertebral bone marrow pathological lesions.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with vertebral lesions Clinically suspected or diagnosed by other modalities as X-ray or CT were included in the study.

Exclusion Criteria:

* Patients with metallic prosthesis which are not MRI compatible .
* patients with previous Vertebral surgery.
* patients with Vertebral Congenital anomalies
* Patients refused the examination.
* Patients who suffer from claustrophobia

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: - All adult patients with various vertebral bone marrow lesions.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of MRI diffusion in differentiation between Various Vertebral bone marrow pathological lesions. . | Baseline
  Primary (main):
  Establishing correlations between DWI findings and laboratory, clinical or histopathological results.

CONTACTS AND LOCATIONS:
Overall Officials: Eman A. Ahmed, Study Director — Professor; Shimaa F. Gad, Study Director — Assistant professor

REFERENCES:
- [Background] Leake RL, Mills MK, Hanrahan CJ. Spinal Marrow Imaging: Clues to Disease. Radiol Clin North Am. 2019 Mar;57(2):359-375. doi: 10.1016/j.rcl.2018.09.008. Epub 2018 Nov 17. PMID 30709475
- [Background] Lin S, Ouyang T, Kanekar S. Imaging of Bone Marrow. Hematol Oncol Clin North Am. 2016 Aug;30(4):945-71. doi: 10.1016/j.hoc.2016.03.012. PMID 27444005
- [Background] Dietrich O, Geith T, Reiser MF, Baur-Melnyk A. Diffusion imaging of the vertebral bone marrow. NMR Biomed. 2017 Mar;30(3). doi: 10.1002/nbm.3333. Epub 2015 Jun 26. PMID 26114411
- [Background] Karampinos DC, Ruschke S, Dieckmeyer M, Diefenbach M, Franz D, Gersing AS, Krug R, Baum T. Quantitative MRI and spectroscopy of bone marrow. J Magn Reson Imaging. 2018 Feb;47(2):332-353. doi: 10.1002/jmri.25769. Epub 2017 Jun 1. PMID 28570033
- [Background] Padhani AR, Koh DM. Diffusion MR imaging for monitoring of treatment response. Magn Reson Imaging Clin N Am. 2011 Feb;19(1):181-209. doi: 10.1016/j.mric.2010.10.004. PMID 21129641